CLINICAL TRIAL: NCT07123311
Title: Implementation and Evaluation of an Internet-Based Stress Management Program for Health Students in the Sfax Region
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sfax (Other)
Responsible Party: Principal Investigator, Ines KHARRAT, PhD Student, University of Sfax
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMS-08-05-1982-63-24
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Depression (Mild or Not Persistent)
Keywords: Mental Health; Stress, Psychological / therapy; Students; Internet
MeSH Terms: conditions — Lymphoma, Follicular; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group, randomized controlled trial with a 1:1 allocation ratio. Participants will be randomly assigned to either an intervention group, which will receive an internet-based stress management program inspired by the validated French program "Je gère mon stress", or to a wait-list control group receiving no intervention during the study period. The study is single-blind (with outcome assessors blinded) and will span 8 weeks, including pre- and post-intervention assessments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe I (Experimental): Participants in the intervention group will receive an email containing their login credentials (username and password) to access the website and actively participate in the scheduled sessions of the program. Upon logging in, they will watch a short introductory video of about five minutes explaining how the program works. They will then answer three follow-up questions to confirm their understanding. If any answers are incorrect, they will be asked to rewatch the video until all questions are correctly answered.
  Next, participants will receive an information letter explaining the requirement to visit the website at least once a week for a minimum of 30 minutes per session, with the option to spend more time or visit more frequently if they wish. After successfully answering the questions, they will be asked to provide informed consent ensuring the security and confidentiality of their personal data before accessing the sessions.
  This initial step is crucial for the success of the p
  Interventions: Behavioral: Online Stress Management Program
- Groupe C (No Intervention): Participants in the control group will receive an email informing them of their assignment. They will have access to the website after 12 weeks. They will be asked to refrain from any stress management activities (such as yoga, meditation, etc.) during this period.

INTERVENTIONS:
Behavioral: Online Stress Management Program — This is an online pilot stress management program tailored for health students, combining cognitive-behavioral therapy and guided mindfulness meditation. Over eight sessions, participants engage with interactive psychoeducation modules, videos, and practical exercises to understand stress and develop coping strategies.
  The sessions cover stress awareness, mindfulness meditation (basic and advanced), breathing techniques, time management using the Eisenhower matrix, and cognitive-behavioral methods to foster positive thinking and problem-solving.
  The final session helps participants create a personalized action plan to integrate learned skills into daily life. Throughout the program, a support group encourages interaction and provides ongoing guidance to enhance well-being and stress management.
  Arms: Groupe I

SUMMARY:
The objective of this experimental study (randomized controlled trial) is to evaluate the effectiveness of an internet-based stress management program, inspired by the French program "Je gère mon stress," among healthcare students in Sfax, Tunisia.

The target population includes all healthcare students over 18 years old, from any field (paramedical, nursing, medicine, etc.), regardless of their baseline level of perceived stress.

The main questions this study aims to answer are:

Does the online program significantly reduce the level of perceived stress (measured using the Perceived Stress Scale - PSS-10)? Does the program have a beneficial impact on symptoms of anxiety and depression (measured with the Hospital Anxiety and Depression Scale - HADS)? Does it improve sleep quality (assessed using the Pittsburgh Sleep Quality Index - PSQI)?

Comparison group:

Researchers will compare the outcomes of the intervention group (who will access the online stress management program for 8 weeks) with those of the control group (waiting list, no initial access), to evaluate the specific effects of the program.

Participants will:

Complete three validated questionnaires (PSS-10, HADS, and PSQI) before and after the intervention; Be invited to follow a weekly series of psychoeducational modules over 8 weeks, including short educational videos, breathing techniques, guided relaxation, and practical exercises, all accessible through a secure web platform; Receive weekly motivational messages to support engagement.

DETAILED DESCRIPTION:
This randomized controlled trial aims to assess the effectiveness of an internet-based stress management program tailored for healthcare students in Sfax, Tunisia. The intervention is an adaptation of the validated French program "Je gère mon stress," redesigned to fit the local sociocultural context.

The study targets healthcare students aged 18 and above, from various disciplines (nursing, physiotherapy, midwifery, anesthesia, etc.), regardless of their baseline perceived stress levels.

Participants in the intervention group will receive access to an 8-week structured online program composed of:

Weekly psychoeducational video capsules (covering stress mechanisms, coping strategies, relaxation techniques, etc.), Guided breathing and relaxation exercises, Simple cognitive-behavioral tools, Time management and lifestyle advice.

All participants will be assessed at baseline (pre-intervention) and post-intervention using three validated instruments:

PSS-10 (Perceived Stress Scale) to evaluate perceived stress, HADS (Hospital Anxiety and Depression Scale) to assess symptoms of anxiety and depression, PSQI (Pittsburgh Sleep Quality Index) to measure sleep quality. A control group will not receive any intervention during the 8-week period but will be offered the program after the study ends (waiting list design). This design allows a fair comparison between groups and ensures ethical access to the intervention.

The program is fully accessible online via a secure platform and requires no in-person attendance. Participants will receive weekly reminders to complete the sessions and questionnaires.

The main outcome is the change in perceived stress levels. Secondary outcomes include changes in anxiety, depression, and sleep quality.

This study contributes to addressing the high psychological burden observed in healthcare students in Tunisia and promotes the use of digital tools for mental health support in academic settings.

ELIGIBILITY:
Inclusion Criteria:

* The target population includes all students enrolled in the second year at the Higher Institute of Nursing Sciences (ISSIS) and the Higher School of Health Sciences and Techniques (ESSTSS) for the 2025-2026 academic year.

Own a smartphone, tablet, or computer. Have internet access. Have an email address. Be willing to be randomized. Have given informed consent to participate in the study. Be available and committed to completing the entire online intervention program and participating in all evaluations.

Exclusion Criteria:

* The study does not have any specific a priori exclusion criteria. However, participants will be excluded from the analysis in the following cases:

Voluntary withdrawal: any participant wishing to stop their participation may do so at any time; Incomplete data: data that do not allow for reliable statistical analysis will be excluded from the final analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Level in Health Students | At baseline (week 0), at the end of the program (week 8), and one month post-intervention (week 12)
  This measure assesses participants' perceived stress intensity before and after the intervention using a validated tool such as the Perceived Stress Scale (PSS). It quantifies changes in stress management and evaluates the program's impact on students' psychological well-being.Follow-up assessment will also be conducted one month after the program ends to evaluate the long-term effects.

SECONDARY OUTCOMES:
Anxiety and Depression Levels (HADS) and Sleep Quality (Pittsburgh Sleep Quality Index) | At baseline (week 0), at the end of the program (week 8), and one month post-intervention (week 12)
  This measure assesses anxiety and depression symptoms using the Hospital Anxiety and Depression Scale (HADS) and evaluates sleep quality through the Pittsburgh Sleep Quality Index (PSQI). These validated tools will track changes in participants' anxiety, depression, and sleep disturbances before and after the intervention, providing a comprehensive view of the program's impact on mental health and well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Rim Masmoudi, Professor in Medicine, Study Director — University of Sfax; Jihen Jdidi, Professor in Medicine, Study Director — University of Sfax
Locations (1):
- Faculties of Sealth Sciences, Sfax, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 6 months after publication of the main results in a peer-reviewed journal.
Access Criteria: Qualified researchers affiliated with academic or health research institutions will be able to access anonymized individual participant data (IPD), the study protocol, and statistical analysis plan upon request. Access will be granted for scientifically valid research purposes, such as meta-analyses or secondary analyses on mental health interventions. Data will be shared via secured email or encrypted file transfer, following the approval of a data use agreement and submission of a research proposal to the principal investigator.